CLINICAL TRIAL: NCT02340078
Title: A Randomized, Multi Center, Double-blind, Active-controlled, Matched Pairs Design Clinical Study to Evaluate the Efficacy and Safety of HA IDF II Plus Versus HA IDF II in Nasolabial Fold Injection
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of YVOIRE Volume Plus Versus YVOIRE Volume in Nasolabial Fold Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LG-HACL011
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2013-11

CONDITIONS: Wrinkles
Keywords: the facial nasolabial fold

STUDY DESIGN:
Intervention Model Description: Split-face design. Subjects were decided by randomization which side of the face would be injected with the test device. According to this randomization result, the other side would be determined to be injected with a comparator. It was determined just by one randomization.
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- HA IDF II (Active Comparator): cross-linked HA filler
  Interventions: Device: HA IDF II
- HA IDF II plus (Experimental): cross-linked HA filler with lidocaine
  Interventions: Device: HA IDF II plus

INTERVENTIONS:
Device: HA IDF II plus
  Arms: HA IDF II plus
Device: HA IDF II
  Arms: HA IDF II

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of HA IDF II plus (with lidocaine) injected in the nasolabial fold compared to HA IDF II (without lidocaine).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 30 and 60
2. Those whose wrinkles in the treatment area (nasolabial fold) correspond to Stage 3 or 4 in the 5-stage Wrinkle Severity Rating Scale (WSRS) symmetrically
3. Those who were informed on the purpose, method, and effect etc. of this study and signed the informed consent form
4. Those who fell under any of the following 3 cases:

   1. Surgically sterile women
   2. Women in menopause over 2 years from the last menstruation, aged at least 45
   3. Among the women meeting neither of a nor b, those who agreed to use at least 2 contraception methods specified below (one of the barrier methods must be included) until 14 days after the last treatment with the investigational device

      * Barrier methods: Condom, diaphragm, cervical cap (pessary), spermicide
      * Hormonal methods: Pills, injection (depot), skin patch, hormonal implant (Implanon), vaginal ring
      * Intrauterine devices (IUDs): Cooper IUD (Loop), hormonal IUD (Mirena)
      * Natural methods: Basic body temperature, ovulation period, coitus interruptus, abstinent

Exclusion Criteria:

1. Those with a skin disease (skin infection, eczema, psoriasis, rosacea, herpes etc.) in the lower 2/3 part of the face in which the wrinkle evaluation may be affected
2. Patients with a malignant tumor recognized medically important and considered as potentially affecting the clinical study
3. Women in pregnancy or lactation
4. Those with the bilirubin level exceeding 1.5 times of the upper limit of normal or the ALT/AST level exceeding 2.5 times of the upper limit of normal
5. Those with the confirmed infection of syphilis or HIV
6. Those who had an anticoagulant therapy or antiplatelet therapy within 2 weeks prior to Visit 1 (screening)
7. Those who used a topical preparation (steroid, retinoid) in the facial area within 4 weeks prior to Visit 2 (randomization )
8. Those who experienced a deep chemical peeling or a procedure judged as potentially affecting the clinical study within 3 months prior to Visit 2 (randomization)
9. Those who experienced a non-permanent filler procedure or a cosmetic surgery in the face within 9 months prior to Visit 2 (randomization)
10. Those who had an implantation procedure with a permanent substance (silicone, PAAG, PMMA, CaHA etc.) in the treatment area (nasolabial fold )
11. Those currently with a streptococcal disease
12. Those with a history of severe allergy or hypersensitivity (anaphylaxis) judged as potentially affecting the clinical study
13. Those with a history of hypertrophic scar or keloid
14. Those with a history of bleeding disorder
15. Those with a hypersensitivity to the investigational device of this clinical study or lidocaine
16. Those who refused to agree not to use a local or systemic pain-relieving agent or other pain-relieving method (e.g.: ice pack) from the midnight of the treatment day with the investigational device through the post-measurement of the last VAS pain scale
17. Those who had participated in another clinical study within 1 month prior to Visit 1 (screening)
18. Those judged by the investigator as ineligible for this clinical study

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: at 2 hospitals in korea, 62 patients. period : Nov 2013~Feb 2015
Pre-assignment Details: spilt-face design. Subjects were decided by randomization which side of the face would be injected with the test device. According to this randomization result, the other side would be determined to be injected with a comparator. It was determined just by one randomization.
Groups:
- Subject Disposition: All Study Participants
Period: Overall Study
Arm/Group | Subject Disposition
Started | 62
Completed | 61
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Demographic Charateristics: Subjects who were included in efficacy evaluation
Arm/Group | Demographic Charateristics
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.39 (7.03)
Sex/Gender, Customized [Number; unit: participants]
  Female | 62
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of the Subjects With at Least 10mm Difference in VAS Pain Scale Scores Within the Subject (VAS of the Control Device - VAS of the Test Device) Immediately After Treatment With the Investigational Devices
Description: The degree of pain was evaluated by VAS (Visual Analog Scale), measuring the length from the left and to the mark by the subject in millimeter (mm) unit.
Time Frame: Visit 2 (week 0, immediately after treatment)
Measure: Number; unit: participants
Groups:
- Subjects With at Least a 10mm Difference in VAS: Subjects with at least a 10mm difference in VAS (HA IDF II - HA IDF II plus)
- Subjects With Below 10mm Difference in VAS: Subjects with below 10mm difference in VAS (HA IDF II - HA IDF II plus)
Arm/Group | Subjects With at Least a 10mm Difference in VAS | Subjects With Below 10mm Difference in VAS
Number analyzed (Participants) | 62 | 62
participants | 59 | 3
Statistical Analysis 1: Comparison: Subjects With at Least a 10mm Difference in VAS vs Subjects With Below 10mm Difference in VAS; Test type: Superiority; Subjects % with difference in VAS ≥ 10mm = 0.9516, 95% CI 2-sided [0.87 to 0.99]

ADVERSE EVENTS:
Groups:
- Safety: Subject who were injected with investigational medical device at least once.
  The 'Serious Adverse Events' and 'Other Adverse Events' described below occured in each subject regardless of the left or right of the injection site, and since all subjects were injected with both test device and comparator, it was not indicated which side the test device was injected.
Arm/Group | Safety
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 3/62
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety (N=62)
Administration Site Conditions (General disorders) | 3 (3) — In detail, 'Injection Site Discomfort' were 3 cases, showing the highest incidence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other